CLINICAL TRIAL: NCT06201234
Title: Phase II Study Evaluating the Addition of Elacestrant, an Oral Selective Estrogen Receptor Degrader (SERD), to Standard-of-care Olaparib in Patients With Hormone Receptor (HR)-Positive, HER2-negative Locally Advanced or Metastatic Breast Cancer With gBRCA1/2 Mutations
Brief Title: Evaluating the Addition of Elacestrant (Oral SERD) to Olaparib (PARP-inhibitor) in Patients With Advanced/Metastatic HR+/HER2- Breast Cancer
Acronym: ELEMENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELEMENT GBG-114
Record Dates: First submitted 2023-12-07; First posted 2024-01-11 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hormone Receptor Positive HER-2 Negative Breast Cancer; Advanced or Metastatic Breast Cancer; BRCA1 Mutation; BRCA2 Mutation
Keywords: Elacestrant; Olaparib; Breast cancer; Metastases; Palliative therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — olaparib; elacestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Olaparib + elacestrant* (Experimental): Treatment will be given until disease progression, unacceptable toxicity, withdrawal of patient´s consent to study participation, or end of study.
  * Together with GnRH analogue in pre- and perimenopausal women, and in men, at least two weeks prior to treatment.
  * Elacestrant tablets 400 mg orally daily
  * Olaparib 600 mg orally daily The protocol provides procedures for specific adverse events requiring dose modifications or delays.
  Interventions: Drug: Olaparib + Elacestrant
- Arm B: Olaparib (Active Comparator): Treatment will be given until disease progression, unacceptable toxicity, withdrawal of patient´s consent to study participation, or end of study.
  • Olaparib 600 mg orally once daily
  The protocol provides procedures for specific adverse events requiring dose modifications or delays.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib + Elacestrant — Olaparib 600 mg orally daily and elacestrant 400 mg orally daily
  Arms: Arm A: Olaparib + elacestrant*
Drug: Olaparib — Olaparib 600 mg orally daily
  Arms: Arm B: Olaparib

SUMMARY:
Trial design:

Phase II, prospective, multi-center, randomized, open label, parallel group study in patients with HR-positive, HER2-negative locally advanced or metastatic breast cancer with gBRCA1/2 mutation, with 2:1 randomization into Arm A (olaparib + elacestrant) or arm B (olaparib). Treatment in either arm will be given until disease progression, unacceptable toxicity, withdrawal of patient´s consent to study participation, or end of study.

Trial population:

Patients with HR-positive, HER2-negative locally advanced or metastatic breast cancer with gBRCA1/2 mutation, with an indication for standard-of-care PARP inhibitor therapy and planned treatment with olaparib, an ECOG performance status of 0-2 and life expectancy of > 6 months, with normal bone marrow and kidney functions and no active or newly diagnosed central nervous system (CNS) metastases or symptomatic metastatic visceral disease at risk of life-threatening complications.

Interventions:

Patients randomized to Arm A will receive 600 mg olaparib daily and 400 mg elacestrant daily, while patients randomized to Arm B will receive 600 mg olaparib daily. Blood tests (hematology, biochemistry) will be performed at the beginning of every cycle, and imaging for tumor assessment (chest and abdominopelvic imaging) as well as QoL assessments will be performed every three months and in case of suspicion of progression/end of study.

DETAILED DESCRIPTION:
Patients with HR-positive, HER2-negative advanced or metastatic breast cancer and gBRCA1/2 mutations have a low progression-free survival (PFS) and represent a patient population with a high unmet need, hence further treatment options should be explored to improve patient outcomes.

Elacestrant is a novel, nonsteroidal, orally bioavailable estrogen receptor antagonist (SERD) that has shown efficacy in heavily pretreated patients with HR-positive, HER2-negative breast cancer, and in those with ESR1 mutations known to confer endocrine resistance, and has thus gained approval in 2023 by the Food and Drug Administration (FDA) and the European Medicines Agency (EMA) for postmenopausal women or adult men with ER-positive, HER2-negative, ESR1-mutated advanced or metastatic breast cancer with disease progression following at least one line of ET.

Olaparib is approved by the EMA for deleterious or suspected deleterious gBRCA-mutated, HER2-negative metastatic BC, based on positive outcomes in the phase III OlympiAD trial which showed improved median PFS, response rates, and less toxicity with olaparib compared to SOC.

The purpose of the proposed study is to investigate if the addition of elacestrant to standard olaparib therapy could potentially lead to an improvement in PFS compared to olaparib alone in patients with HR-positive, HER2-negative locally advanced or metastatic breast cancer with gBRCA1/2 mutations.

ELEMENT is a phase II, prospective, multi-center, randomized, open label, parallel group study in patients with HR-positive, HER2-negative locally advanced or metastatic breast cancer with gBRCA1/2 mutation, with 2:1 randomization into Arm A (olaparib + elacestrant) or arm B (olaparib). Treatment in either arm will be given until disease progression, unacceptable toxicity, withdrawal of patient´s consent to study participation, or end of study.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for study participation only if they comply with the following criteria:

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for scheduled visit, the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
2. Female or male patients.
3. Age at study entry of at least 18 years.
4. Locally advanced or metastatic breast cancer that is HR-positive (ER and/or PgR ≥ 10% of stained cells at IHC) and HER2-negative (IHC 0 or 1+, or 2+ and ISH negative according to ASCO/CAP guidelines).
5. Patients with deleterious or suspected deleterious gBRCA1/2 mutation detected upon local testing.
6. Willingness and ability to provide archived formalin fixed paraffin embedded tissue (FFPE) block or a partial block from archived tumor or metastasis.
7. Indication for standard-of-care PARP inhibitor therapy and planned treatment with olaparib.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
9. Resolution of all acute toxic effects of prior anti-cancer therapy including endocrine therapy or surgical procedures to NCI CTCAE version 5.0 grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
10. Life-expectancy > 6 months.
11. For female patients: patients of childbearing potential (defined as not post-menopausal and not permanently sterile [latter defined as having undergone hysterectomy, bilateral salpingectomy, or bilateral oophorectomy]) require a negative serum or urinary pregnancy test within 72 hours before starting treatment in this study (in this case, patients need to use highly effective non-hormonal contraceptive methods as specified in the protocol).

For male patients: during the intervention period and for at least 120 days after the last dose of elacestrant, patients should refrain from heterosexual intercourse or use a condom (and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak), and they should refrain from donating sperm.

Exclusion Criteria:

Patients will be ineligible for study participation if they fulfill any of the following criteria:

1. Known hypersensitivity reaction to one of the compounds, excipients, or substances used in this protocol.
2. Active or newly diagnosed CNS metastases, including leptomeningeal carcinomatosis, carcinomatous meningitis, or radiographic signs of CNS hemorrhage. Note: Patients with stable brain metastases are allowed. Radiotherapeutic treatment must be completed 1 week before planned day 1 of study therapy.
3. Presence of symptomatic metastatic visceral disease that are at risk of life-threatening complications in the short term, including but not confined to massive uncontrolled effusions (peritoneal, pleural, pericardial), pulmonary lymphangitis, or fulminant liver involvement.
4. Inadequate organ function prior to enrolment including:

   * Hemoglobin < 9 g/dL (< 5.6 mmol/L)
   * Absolute neutrophil count (ANC) < 1500/mm³ (< 1.5 x 109/L)
   * Platelets < 100,000/mm³ (< 100 x 109/L)
   * Alanine aminotransferase (ALT/SGPT) and/or aspartate aminotransferase (AST/SGOT) > 3 x upper normal limits (ULN). If the patient has liver metastases, ALT and AST should not be ≥ 5 x ULN.
   * Alkaline phosphatase (ALP) > 2.5 x ULN
   * Total serum bilirubin > 1.5 x ULN (exception: patients with Gilbert's syndrome permitted up to ≤ 3 x ULN)
   * Serum creatinine > 1.5 x ULN or estimated creatinine clearance < 50 mL/min as calculated using the standard method for the institution.
5. Existing contraindication against the use of the elacestrant or olaparib.
6. Prior treatment with PARP inhibitors.
7. Female patients: pregnancy or lactation at the time of randomization or intention to become pregnant during the study and for a predefined period after the end of treatment (as described in protocol).

   Male patients: intention to get a child during the study and for a predefined period after the end of treatment (as described in protocol).

   According to the treatment received during the study, required contraception timelines for female and male patients are described in the study protocol.
8. Any of the following within 6 months prior to enrolment: myocardial infarction, severe/unstable angina, ongoing grade ≥ 2 cardiac dysrhythmias, prolonged QT corrected by Fridericia's formula (QTcF) grade ≥ 2, uncontrolled atrial fibrillation of any grade, coronary/peripheral artery bypass graft, heart failure of New York Heart Association (NYHA) Class II or greater, or cerebrovascular accident including transient ischemic attack.
9. Uncontrolled hypertension at the time of screening (systolic BP > 140 mmHg or diastolic BP > 90 mmHg that has not been adequately treated or controlled).
10. Active and current anticoagulation for treatment purposes of thrombotic events occurring < 6 months before enrolment is not allowed (prophylactic anticoagulation, however, is acceptable). Treatment with an anticoagulant for a thrombotic event occurring > 6 months before enrolment, or for an otherwise stable and allowed medical condition (e.g., well controlled atrial fibrillation) is acceptable, provided dose and coagulation parameters (as defined by local standard of care) are stable for at least 28 days prior to the first dose of study drug.
11. Known difficulty in tolerating oral medications or conditions which would impair absorption of oral medications such as: uncontrolled nausea or vomiting (i.e., CTCAE ≥ grade 3 despite antiemetic therapy), ongoing gastrointestinal obstruction/motility disorder, malabsorption syndrome, or prior gastric bypass.
12. History of endometrial intraepithelial neoplasia in patients who have not undergone a hysterectomy.
13. Malignant disease other than breast cancer, active or being disease-free for less than 5 years (except carcinoma in situ of the cervix, DCIS, and non-melanomatous skin cancer adequately treated).
14. Uncontrolled significant active infections including HBV, HCV, and/or HIV. Patients with a positive hepatitis B surface antigen result or a positive hepatitis C antibody test result at screening or within 3 months before first dose of study treatment are excluded, except for the following:

    * Participants with positive anti-HBs antibody titer and confirmatory negative hepatitis B DNA polymerase chain reaction.
    * Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled only if they have both completed curative therapy and have a hepatitis C viral load < quantifiable limit.
15. Any severe, acute, uncontrolled, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational or non-investigational products administration, or may interfere with the interpretation of study results, and, in the judgment of the investigator, would make the patient inappropriate for entry into this study. Moreover, patients who, by virtue of an order issued by judicial or administrative authorities, are committed to an institution or those who cannot take part in clinical trials are excluded from this study.
16. History of significant neurological or psychiatric disorders including psychotic disorders, dementia, or seizures that would prohibit the understanding and giving of informed consent.
17. Unable or unwilling to avoid medications, supplements (e.g., St. John's wort), or foods (e.g., grapefruit, pomegranate, pomelos, star fruit, Seville oranges and their juices) that are moderate/strong inhibitors or inducers of CYP3A4 activity. Participation will be allowed if the medication, supplements, or foods are discontinued for at least 14 days prior to study entry and for the duration of the study.
18. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
19. Receipt of live attenuated vaccination within 30 days prior to study entry. COVID-19 vaccines that do not contain live viruses are allowed (at least one week prior to study entry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | PFS is defined as the time from randomization to first progression as assessed by the investigator, or death, whichever occurs first, assessed up to 48 months.
  PFS, investigator-assessed. To evaluate the impact on PFS of elacestrant with olaparib compared to olaparib alone in patients with hormone receptor (HR)-positive, HER2-negative locally advanced or metastatic breast cancer with gBRCA1/2 mutations.

SECONDARY OUTCOMES:
Time-to-treatment failure (TTF) | TTF is defined as time from randomization to discontinuation of treatment due to disease progression, treatment toxicity, patient´s preference, or death, assessed up to 48 months.
  To compare TTF between treatment arms (i.e., elacestrant + olaparib vs. olaparib).
Overall survival (OS) | OS is defined as the time from randomization to death due to any reason, assessed up to 48 months.
  To compare OS between treatment arms.
Patient reported outcome (PRO) in the form of quality of life (QoL) assessment | At baseline, day 1 of cycle 2 (each cycle is 28 days), every 3 months starting from treatment start, and at end of treatment (an average of 12 months per patient).
  To assess and compare patient reported breast cancer-specific QoL as measured by FACT-ES questionnaire.
PFS in stratified and exploratory subgroups | PFS is defined as the time from randomization to first progression as assessed by the investigator, or death, whichever occurs first, assessed up to 48 months.
  To compare PFS in the stratified subgroups: pre-treatment chemotherapy in the metastatic setting yes vs. no.
  To compare PFS in the exploratory subgroups specified in the protocol.
TTF in the stratified subgroups | TTF is defined as time from randomization to discontinuation of treatment due to disease progression, treatment toxicity, patient´s preference, or death, assessed up to 48 months.
  To compare TTF in the stratified subgroups: pre-treatment chemotherapy in the metastatic setting yes vs. no.
  To compare TTF in the exploratory subgroups specified in the protocol.
OS in the stratified subgroups | OS is defined as the time from randomization to death due to any reason, assessed up to 48 months.
  To compare OS in the stratified subgroups: pre-treatment chemotherapy in the metastatic setting yes vs. no.
  To compare OS in the exploratory subgroups specified in the protocol.
Overall response rate (ORR) | ORR is defined as the percentage of patients who have achieved either a confirmed complete response or partial response, assessed up to 48 months.
  To compare ORR between treatment arms.
Clinical benefit rate (CBR) | CBR is defined as the percentage of patients who have achieved either a confirmed complete response or partial response, or stable disease for at least 24 weeks from randomization.
  To compare the CBR between treatment arms.
Numbers and types of adverse events as assessed by CTCAE v5.0 | During treatment phase, an average of 12 months per patient.
  To assess and compare safety between treatment arms (frequency and severity of AEs graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0).
Compliance between treatment arms as assessed by treatment delays, reductions, and interruptions | During treatment phase, an average of 12 months per patient.
  Frequencies of patients whose treatment had to be reduced, delayed, interrupted, or prematurely discontinued will be reported for both arms, together with reasons for such modifications, and comparisons between the two arms will be conducted with the χ2-test with continuity correction.

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, MD, PhD, Study Chair — Prof., MD ASCO, ESGO, ESMO, DKG, DGGG, AGO, DGS, BIG, BCIRG, St. Gallen Faculty Member, SABCS Faculty member
Locations (36):
- Germany (36):
  - Vinzenz Von Paul Kliniken gGmbH - Marienhospital, Stuttgart, Baden-Wurttemberg
  - University Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - Rems-Murr-Klinik-Winnenden, Winnenden, Baden-Wurttemberg
  - GRN Klinik Weinheim, Weinheim, Baden-Württembergs
  - Hämatologie-Onkologie im Zentrum MVZ GmbH, Augsburg, Bavaria
  - Klinikum Bayreuth, Bayreuth, Bavaria
  - Schwerpunktpraxis der Gynäkologie und Onkologie, Fürstenwalde, Brandenburg
  - Agaplesion Frankfurter Diakonie Kliniken gGmbH, Frankfurt am Main, Hesse
  - Klinikum der J. W. Goethe Universität, Frankfurt am Main, Hesse
  - Klinikum Kassel GmbH - Frauenklinik, Kassel, Hesse
  - St. Josefs-Hospital, Gynäkologie und Geburtshilfe, Wiesbaden, Hesse
  - Studien GbR Braunschweig, Braunschweig, Lower Saxony
  - MVZ Onkologische Kooperation Harz GbR, Goslar, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinik Köln, Cologne, North Rhine-Westphalia
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Zentrum für Gynäkologische Onkologie am MVZ Medical Center Düsseldorf GmbH, Düsseldorf, North Rhine-Westphalia
  - KEM Kliniken Essen-Mitte GmbH, Essen, North Rhine-Westphalia
  - Marienhospital Witten, Witten, North Rhine-Westphalia
  - Helios Universitätsklinikum Wuppertal, Wuppertal, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Mainz, Rhineland-Palatinate
  - Institut für Versorgungsforschung Mayen, Mayen, Rhineland-Palatinate
  - Caritas Traegergesellschaft Saarbruecken mbH (CTS), Saarbrücken, Saarland
  - University Hospital Carl Gustav Carus, Dresden, Saxony
  - Gemeinschaftspraxis Dr.Illmer, Dr. Wolf, Dr. Jacobasch, Dr. Freiberg-Richter, Dresden, Saxony
  - Universität Leipzig, Leipzig, Saxony
  - MediOnko-Institut GbR, Berlin, State of Berlin
  - Das Brust Zentrum - Die Frauenärzte, Berlin, State of Berlin
  - Marienhospital Bottrop gGmbH, Bottrop
  - Universitätsklinikum Essen - Klinik für Frauenheilkunde und Geburtshilfe, Essen
  - National Center for Tumor Diseases Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes - Frauenklinik, Homburg
  - Rotkreuzklinikum München, München
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Robert Bosch Gesellschaft fuer medizinische Forschung mbH, Stuttgart
  - Klinikum Worms, Worms

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article can be made available after final analysis and publication of all secondary efficacy endpoints.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning after final analysis and publication of all secondary efficacy endpoints; no end date.
Access Criteria: Who: Researchers who provide translational research proposals. Proposals should be approved by the GBG scientific board.
  What: Individual participant data that underlie the results reported in this article, after final analysis and publication of all secondary efficacy endpoints.
  How: Proposal forms should be requested from trafo@gbg.de; once the application has been approved and a data transfer agreement has been signed, researchers will be given access to the data.

REFERENCES:
- [Background] Bidard FC, Kaklamani VG, Neven P, Streich G, Montero AJ, Forget F, Mouret-Reynier MA, Sohn JH, Taylor D, Harnden KK, Khong H, Kocsis J, Dalenc F, Dillon PM, Babu S, Waters S, Deleu I, Garcia Saenz JA, Bria E, Cazzaniga M, Lu J, Aftimos P, Cortes J, Liu S, Tonini G, Laurent D, Habboubi N, Conlan MG, Bardia A. Elacestrant (oral selective estrogen receptor degrader) Versus Standard Endocrine Therapy for Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Results From the Randomized Phase III EMERALD Trial. J Clin Oncol. 2022 Oct 1;40(28):3246-3256. doi: 10.1200/JCO.22.00338. Epub 2022 May 18. Erratum In: J Clin Oncol. 2023 Aug 10;41(23):3962. doi: 10.1200/JCO.23.01239. PMID 35584336
- [Background] Robson M, Im SA, Senkus E, Xu B, Domchek SM, Masuda N, Delaloge S, Li W, Tung N, Armstrong A, Wu W, Goessl C, Runswick S, Conte P. Olaparib for Metastatic Breast Cancer in Patients with a Germline BRCA Mutation. N Engl J Med. 2017 Aug 10;377(6):523-533. doi: 10.1056/NEJMoa1706450. Epub 2017 Jun 4. PMID 28578601
- [Background] Gelmon KA, Fasching PA, Couch FJ, Balmana J, Delaloge S, Labidi-Galy I, Bennett J, McCutcheon S, Walker G, O'Shaughnessy J; Collaborating Investigators. Clinical effectiveness of olaparib monotherapy in germline BRCA-mutated, HER2-negative metastatic breast cancer in a real-world setting: phase IIIb LUCY interim analysis. Eur J Cancer. 2021 Jul;152:68-77. doi: 10.1016/j.ejca.2021.03.029. Epub 2021 Jun 1. PMID 34087573
- [Background] Bardia A, Kaklamani V, Wilks S, Weise A, Richards D, Harb W, Osborne C, Wesolowski R, Karuturi M, Conkling P, Bagley RG, Wang Y, Conlan MG, Kabos P. Phase I Study of Elacestrant (RAD1901), a Novel Selective Estrogen Receptor Degrader, in ER-Positive, HER2-Negative Advanced Breast Cancer. J Clin Oncol. 2021 Apr 20;39(12):1360-1370. doi: 10.1200/JCO.20.02272. Epub 2021 Jan 29. PMID 33513026
- See also: Website of German Breast Group — http://gbg.de